CLINICAL TRIAL: NCT07133984
Title: STICH3C Cardiac Magnetic Resonance (CMR) Observational Study (STICOS)
Brief Title: STICH3C Cardiac Magnetic Resonance Observational Study
Acronym: STICOS
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 23-09026465; 1R01HL170566-01 (NIH)
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Left Ventricle Systolic Dysfunction; Multivessel Coronary Artery Disease
Keywords: iLVSD; CAD; Cardiac MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with iLVSD and CAD undergoing revascularization.: Eligible patients will be approached by study team before PCI or CABG for consent to participate in the study. For patients in whom the treating physicians have requested or will request pre-procedure CMR for clinical reasons, consent to collect long-term clinical data will be requested. Eligible patients who meet inclusion criteria in whom clinical CMR is not planned, will be asked to undergo preoperative CMR with or without postoperative CMR and to be followed up for research purposes.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging — Cardiac MRI, also known as cardiac magnetic resonance imaging, is a non-invasive imaging technique that uses strong magnetic fields and radio waves to produce detailed pictures of the heart and its surrounding structures
  Other Names: CMR

SUMMARY:
STICOS will test the hypothesis that residual jeopardized myocardium, late gadolinium enhancement, and non-ischemic substrate after revascularization is associated with postoperative adverse cardiovascular events such as heart failure , readmission, or death.

This study will look at whether certain heart tissue abnormalities seen on MRI scans can help predict serious health problems after heart procedures like stents or bypass surgery.

DETAILED DESCRIPTION:
iLVSD (ischemic left ventricular dysfunction) is a leading cause of heart failure (HF) and death. It is widely treated via coronary revascularization despite limited understanding of determinants of revascularization response.

"Viability" imaging (to differentiate infarcted from salvageable myocardium) has been widely touted as an effective means to predict revascularization response. However prior multicenter trials have derived negative conclusions using heterogenous data with respect to both image modality and analysis.

Data by our investigators and others indicate that infarct transmurality on CMR strongly impacts remodeling and prognosis after coronary revascularization. The investigators have also developed new methods (dark-blood late gadolinium enhancement-CMR) to assess infarction and shown ischemia (hypoperfusion) and non-ischemic substrate on CMR to strongly impact LV remodeling. Despite conceptual rationale, utility of multiparametric CMR to elucidate mechanism and determinants of remodeling and differential outcomes after percutaneous and surgical revascularization of iLVSD has yet to be tested.

This prospective study will test the hypothesis that residual jeopardized (viable but hypoperfused) myocardium, LGE, and non-ischemic substrate after coronary revascularization (by PCI or CABG) is associated with postoperative adverse cardiovascular events

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years old
2. LVEF ≤ 40% (quantified by echo, single-photon emission computed tomography [SPECT], or CMR within 2 months of enrollment)
3. Prognostically important CAD: either multivessel CAD (triple vessel or double vessel CAD including left anterior descendant artery (LAD), significant coronary stenosis defined as ≥ 70% based on coronary angiography, fractional flow reserve (FFR) ≤ 0.80 or instantaneous wave-free ratio (iFR) ≤ 0.89) or left main disease (+/- other CAD) for which significant stenosis defined as > 50% based on coronary angiography, intravascular ultrasound (IVUS) minimum luminal area [MLA] value ≤ 6.0 mm2 (< 4.5 mm2 Asian descent), or equivalent optical coherence tomography (OCT) measurements.
4. Planned CABG or PCI within 3 months

Exclusion Criteria:

1. Concomitant valve disease or other condition (e.g., LV aneurysm) requiring surgical repair or replacement
2. Contraindication to CMR (i.e. magnetically activated materials), gadolinium, regadenoson/adenosine/dipyridamole
3. Active neoplasm and/or severe end-organ dysfunction with expected life expectancy less than 5 years.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with iLVSD and multivessel coronary artery disease (CAD) undergoing revascularization (PCI or CABG)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac Magnetic Resonance Imaging (CMR) Indices | 5 years
  The primary objective of this study is to relate Cardiac Magnetic Resonance Imaging (CMR) (infarction, perfusion, and nonischemic substrate) after iLVSD revascularization with long-term outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Gaudino, MD, PhD, MSCE, FEBCTS, FACC, Principal Investigator — Weill Medical College of Cornell University
Locations (9):
- United States (3):
  - NewYork-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - New York Presbyterian - Queens, Flushing, New York
  - Weill Cornell Medicine/NewYork Presbyterian Hospital, New York, New York
- MU Vienna Austria, Vienna, Austria
- Canada (3):
  - Libin Cardiovascular Institute, Calgary, Alberta
  - Universite Laval Quebec (CRIUCPQ) Canada, Québec
  - Sunnybrook Health Sciences Centre, Toronto
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, China
- Dedinje Cardiovascular Institute, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided